CLINICAL TRIAL: NCT06024694
Title: Retrospective Multicenter International Study on Prognostic Factors, Management And Outcome Of Primary Mediastinal Large B-Cell Lymphoma (PMLBCL) Patients With Central Nervous System (CNS) Involvement
Brief Title: Primary Mediastinal Large B-cell Lymphoma With CNS Involvement
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrés José Maria Ferreri, Lymphoma Unit Director, IRCCS San Raffaele
Other Study IDs: OSR PMLBCL SNC+; NCT05856708 (obsolete NCT alias)
Record Dates: First submitted 2022-08-24; First posted 2023-09-06 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Primary Mediastinal Large B-cell Lymphoma (PMBCL)
Keywords: CNS; PMLBCL

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients diagnosed with PMLBL: Patients whose diagnosis met the histological criteria of PMLBL according WHO classification with a diagnosis of CNS involvement at relapse/progression

SUMMARY:
This is a retrospective, multicenter study focused on patients with a known diagnosis of PMLBCL which experienced a CNS relapse during the course of their disease to obtain information about the clinical characteristics, the management at diagnosis and at each relapses , and the outcome of these cases. The aim of the study is to put together the large International series on CNS+ PMLBCL data, coming from 6 different countries , on clinical factors, anti-lymphoma therapy administered alone or concomitant with CNS prophylaxis , the information about the site of re biopsy when available , the dose intensity of lymphoma therapy received at relapse and the outcome of patients.

Both patients treated in routine practice or within clinical trials will be considered. Moreover to better characterized the pathological features of this rare entity a central pathological review of the initial diagnosis and when available of for histological confirmed relapse will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of Primary Mediastinal Large B Cell Lymphoma (PMLBCL) according WHO Classification
* Had a recurrence/progression with Central Nervous System (CNS) involvement
* Availability of details on clinical presentation, treatment details and outcome
* Availability of details on pathological data for central review
* Age ≥18 years

Exclusion Criteria

* Patients with CNS lymphoma other than PMLBCL subtype

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients whose diagnosis met the histological criteria of PMLBL according WHO classification with a diagnosis of CNS involvement at relapse/progression.
  Patients eligible to the study will be retrospectively identified by the site researches by interrogating the local site sources.
  Availability of local pathological report at time of diagnosis and restaging will be considered for eligibility.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2027-06-10 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics 1 | 2 YEARS
  to describe the PMLBCL characteristics at diagnosis and at CNS relapse ( first relapse or second and subsequent recurrences) and the treatment received to describe the median time to CNS relapse to define prognostic factors of outcome of CNS relapse in PMLBCL patients
Clinical characteristics 2 | 2 YEARS
  to correlate treatment strategy with survival end-points
Clinical characteristics 3 | 2 YEARS
  to evaluate the Progression Free Survical ( PFS) after CNS events
Clinical characteristics 4 | 2 YEARS
  to evaluate Overall Survival ( OS) after CNS relapse to centra! pathological reviewed the initial diagnosis and the relapse and to correlate biological and molecular factors with CNS recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cazals-Hatem D, Lepage E, Brice P, Ferrant A, d'Agay MF, Baumelou E, Briere J, Blanc M, Gaulard P, Biron P, Schlaifer D, Diebold J, Audouin J. Primary mediastinal large B-cell lymphoma. A clinicopathologic study of 141 cases compared with 916 nonmediastinal large B-cell lymphomas, a GELA ("Groupe d'Etude des Lymphomes de l'Adulte") study. Am J Surg Pathol. 1996 Jul;20(7):877-88. doi: 10.1097/00000478-199607000-00012. PMID 8669537
- [Background] Falini B, Venturi S, Martelli M, Santucci A, Pileri S, Pescarmona E, Giovannini M, Mazza P, Martelli MF, Pasqualucci L, et al. Mediastinal large B-cell lymphoma: clinical and immunohistological findings in 18 patients treated with different third-generation regimens. Br J Haematol. 1995 Apr;89(4):780-9. doi: 10.1111/j.1365-2141.1995.tb08415.x. PMID 7539625
- [Background] Swerdlow SH, Campo E, Pileri SA, Harris NL, Stein H, Siebert R, Advani R, Ghielmini M, Salles GA, Zelenetz AD, Jaffe ES. The 2016 revision of the World Health Organization classification of lymphoid neoplasms. Blood. 2016 May 19;127(20):2375-90. doi: 10.1182/blood-2016-01-643569. Epub 2016 Mar 15. PMID 26980727
- [Background] Bishop PC, Wilson WH, Pearson D, Janik J, Jaffe ES, Elwood PC. CNS involvement in primary mediastinal large B-cell lymphoma. J Clin Oncol. 1999 Aug;17(8):2479-85. doi: 10.1200/JCO.1999.17.8.2479. PMID 10561312
- [Background] Zinzani PL, Martelli M, Bertini M, Gianni AM, Devizzi L, Federico M, Pangalis G, Michels J, Zucca E, Cantonetti M, Cortelazzo S, Wotherspoon A, Ferreri AJ, Zaja F, Lauria F, De Renzo A, Liberati MA, Falini B, Balzarotti M, Calderoni A, Zaccaria A, Gentilini P, Fattori PP, Pavone E, Angelopoulou MK, Alinari L, Brugiatelli M, Di Renzo N, Bonifazi F, Pileri SA, Cavalli F; International Extranodal Lymphoma Study Group (IELSG). Induction chemotherapy strategies for primary mediastinal large B-cell lymphoma with sclerosis: a retrospective multinational study on 426 previously untreated patients. Haematologica. 2002 Dec;87(12):1258-64. PMID 12495899
- [Background] Martelli M, Ferreri A, Di Rocco A, Ansuinelli M, Johnson PWM. Primary mediastinal large B-cell lymphoma. Crit Rev Oncol Hematol. 2017 May;113:318-327. doi: 10.1016/j.critrevonc.2017.01.009. Epub 2017 Jan 21. PMID 28318892
- [Background] Aoki T, Izutsu K, Suzuki R, Nakaseko C, Arima H, Shimada K, Tomita A, Sasaki M, Takizawa J, Mitani K, Igarashi T, Maeda Y, Fukuhara N, Ishida F, Niitsu N, Ohmachi K, Takasaki H, Nakamura N, Kinoshita T, Nakamura S, Ogura M. Prognostic significance of pleural or pericardial effusion and the implication of optimal treatment in primary mediastinal large B-cell lymphoma: a multicenter retrospective study in Japan. Haematologica. 2014 Dec;99(12):1817-25. doi: 10.3324/haematol.2014.111203. Epub 2014 Sep 12. PMID 25216682